CLINICAL TRIAL: NCT01134146
Title: A Phase I Study of Intensity Modulated Radiotherapy (IMRT) for Malignant Pleural Mesothelioma After Radical Pleurectomy/Decortication (PD)
Brief Title: Radical Pleurectomy/Decortication (PD) and Intensity Modulated Radiotherapy (IMRT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0057; NCI-2011-02080 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer; Mesothelioma
Keywords: Intensity Modulated Radiotherapy; IMRT; Malignant Pleural Mesothelioma; Radical Pleurectomy; Decortication; PD; pleurectomy; lung surgery; pleura
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma; Mesothelioma, Malignant | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensity Modulated Radiation Therapy (IMRT) (Experimental): Intensity Modulated Radiation Therapy (IMRT) Delivery of whole-pleura radiation doses beginning with 1) 45 Gy to low-risk region and 60-66 Gy to high-risk region; then 2) the same dosing regimen as above with a third dosing level, 50 Gy to an intermediate-dosing region. Every weekday (Monday-Friday) for up to 5 weeks, lasting about 45-60 minutes.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT — Delivery of whole-pleura radiation doses beginning with 1) 45 Gy to low-risk region and 60-66 Gy to high-risk region; then 2) the same dosing regimen as above with a third dosing level, 50 Gy to an intermediate-dosing region. Every weekday (Monday-Friday) for up to 5 weeks, lasting about 45-60 minutes.
  Other Names: Intensity modulated radiation therapy

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of radiation that can be given to directly to the pleura (the outer lining of the lungs) using intensity modulated radiation therapy (IMRT) in patients with MM who have had a pleurectomy.

DETAILED DESCRIPTION:
IMRT:

IMRT is a technique to deliver radiation that allows the radiation beam to be shaped around the target area.

Radiation Dose Levels:

If you are found to be eligible to take part in this study, you will be assigned to receive one of two doses of radiation therapy based on when you joined the study. If the first dose is tolerated well by the first group of participants in this study, then the next group of participants will receive the second, higher dose of radiation.

Practice Visit:

You will have a practice radiation visit about 6-14 weeks after your surgery. At this visit, you will have a computed tomography (CT) scan that will be used by the study staff to target where you will receive the IMRT.

A mold will also be made around your body and marks will be made on your skin to help position your body correctly for the IMRT. This practice visit should take about 1-2 hours.

IMRT Visits:

Two (2) weeks after the practice radiation visit, you will begin receiving IMRT. At each visit, you will lie down in the mold of your body that was made at the practice visit and you will be lined up for the IMRT using the marks made at the practice visit. The IMRT will then be delivered. You will receive IMRT every weekday (Monday-Friday) for up to 5 weeks. These visits should last about 45-60 minutes.

Study Visits:

The following tests and procedures will be performed 1 time every week for up to 5 weeks while you are on study:

* You will have a physical and skin exam.
* You will have lung function tests.

You will also have a chest x-ray and a four-dimensional (4D) CT scan to check the status of the disease during the last week that you are receiving IMRT. A 4D CT scan is performed just like a CT scan, but during the 4D CT scan, a small black box (about the size of a deck of cards) will be placed on your abdomen. This box will allow more views of the tumor to be seen during the scan by the study staff.

Length of Study:

You may receive IMRT for up to 5 weeks. The IMRT will be stopped early if the disease gets worse or intolerable side effects occur.

Follow-up Visits:

One (1) month after your last dose of IMRT, you will have a chest x-ray, lung function tests, 4D CT scan and a physical exam. The chest x-ray and CT scan will be performed to check the status of the disease.

Two (2) months after your last dose of IMRT, you will have a chest x-ray and a physical exam.

Three (3) months after your last dose of IMRT, you will have a chest x-ray, lung function tests, a physical exam, a 4D CT scan and a regular CT scan of your chest. The chest x-ray and CT scans will be performed to check the status of the disease.

Long-term Follow-up:

Every 3 months for 2 years, every 6 months for the next 3 years, and 1 time every year after that, you will have lung function tests, a physical exam, and alternating CT and positron emission tomography (PET) scans to check the status of the disease. This means that if you have a CT scan at one visit, you will have a PET scan at the next visit, or vice versa.

This is an investigational study. IMRT given directly to the pleura in patients with MM after a pleurectomy is currently being used for research purposes only.

Up to 22 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have undergone radical pleurectomy/decortication and will be enrolled after surgery.
2. Patients must have had a CT/PET scan prior to surgery
3. Patients will have baseline pulmonary function tests and a quantitative V/Q scan prior to radiation therapy, and then pulmonary function tests one month and three months after the completion of radiation. To be conservative, we will assume that the ipsilateral lung will be nonfunctional after radiation treatment. Therefore, our inclusion criteria for baseline pulmonary function tests are very similar to those that we require prior to an extrapleural pneumonectomy, and are as follows:
4. FEV1 >/= 30% of predicted postoperative (ppoFEV1) (as if the patient underwent a pneumonectomy) based on the following formula using the quantitative V/Q scan: - Predicted post-resection FEV1 = FEV1 x % perfusion to uninvolved lung from the quantitative V/Q scan report.
5. DLCO > 35% predicted
6. Patients must be able to lie flat for the duration of the treatment planning sessions and treatment.
7. Patients must be adequately recovered from surgery and prepared to begin radiation therapy 18 weeks after pleurectomy/decortication. We anticipate that most patients will be ready for radiation simulation between 8-16 weeks after surgery.
8. Patients who have received induction chemotherapy will be included in the study.
9. **Note that 2- 6 represent standard criteria for the delivery of radiation therapy after pleurectomy/decortication, and are not novel criteria for the purposes of this protocol.
10. Age >/= 18.
11. All women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months [i.e., who has had menses at any time in the preceding 12 consecutive months]) and male participants must practice effective contraception (abstinence, oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study.
12. Calculated glomerular filtration rate of 80 mL/min/1.73m^2 with at least 40% of renal contribution from the kidney contralateral to the treated hemithorax, as demonstrated by a pre-radiation renal scan.

Exclusion Criteria:

1. Patients having previous radiation therapy to the low neck, thorax or upper abdomen, unless the previous radiation therapy is clearly out of the current radiation field, as determined by the treating physician
2. Patients with metastatic disease.
3. Patients with any of the following conditions: 1) concomitant malignancies other than squamous cell or basal cell carcinoma of the skin, 2) Carcinoma in situ of the cervix, 3) Uncontrolled acute congestive heart failure defined by New York Heart Association Class III or IV. 4) Patients that have NCCN classified low-risk prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05-27 (Actual); Primary Completion 2017-07-09 (Actual); Study Completion 2017-07-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of IMRT after radical pleurectomy/decortication (PD) | 3 Months
  MTD by assessing the toxicity of two different whole-pleura radiation doses.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gomez, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org